CLINICAL TRIAL: NCT05502562
Title: A Multicentre, Prospective, Non-interventional Single-arm Study Investigating Clinical Parameters Associated With the Initiation of Once-daily Oral Semaglutide in a Real-world Adult Population With Type 2 Diabetes in India
Brief Title: A Research Study to Understand How Oral Semaglutide Works in People With Type 2 Diabetes in India
Acronym: PIONEER REAL
Status: Completed | Type: Observational
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Other Study IDs: NN9924-4960; U1111-1270-0826 (Other: World Health Organization (WHO))
Record Dates: First submitted 2022-08-14; First posted 2022-08-16 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — semaglutide

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Participants with type 2 diabetes: Adult participants with type 2 diabetes and naive to injectable glucose-lowering treatment.
  Interventions: Drug: Oral semaglutide

INTERVENTIONS:
Drug: Oral semaglutide — Participants will be treated with commercially available oral semaglutide according to local label and to routine clinical practice at the discretion of the treating physician. The decision to initiate treatment with commercially available oral semaglutide has been made by the patient/Legally Acceptable Representative (LAR) and the treating physician based on local label before and independently from the decision to include the participant in this study.

SUMMARY:
The purpose of the study is to look at the change in blood sugar levels in participants with type 2 diabetes who start using oral semaglutide. Participants will get oral semaglutide as prescribed to them by the study doctor. The study will last for about 8-11 months (34-44 weeks). Participants will be asked to complete a questionnaire about how they take oral semaglutide tablets. Participants will complete this questionnaire during the normal scheduled visit with the doctor and will be asked questions about their health and their diabetes treatment and lab tests as part of their normal doctor's appointment.

ELIGIBILITY:
Inclusion Criteria:

* Signed consent obtained before any study-related activities (study-related activities are any procedure related to recording of data according to the protocol).
* Diagnosed with type 2 diabetes (T2D).
* The decision to initiate treatment with commercially available oral semaglutide has been made by the patient/Legally Acceptable Representative (LAR) and the treating physician based on local label before and independently from the decision to include the patient in this study.
* Male or female, age above or equal to 18 years at the time of signing informed consent.
* Available glycated haemoglobin A1c (HbA1c) value less than or equal to (<=) 90 days prior to the 'Informed Consent and Treatment Initiation visit' (V1) or HbA1c measurement taken in relation with the 'Informed Consent and Treatment Initiation visit' (V1) if in line with local clinical practice.
* Treatment naive to injectable glucose-lowering drug(s). An exception is short-term insulin treatment for acute illness for a total of less than or equal to (<=) 14 days.

Exclusion Criteria:

* Previous participation in this study. Participation is defined as having given informed consent in this study.
* Any prior or current use of oral semaglutide.
* Hypersensitivity to oral semaglutide or to any of the excipients.
* Treatment with any investigational drug within 30 days prior to signing of informed consent.
* Participation in any clinical trial of an approved or non-approved investigational medicinal product within 30 days prior to signing of informed consent.
* Mental incapacity, unwillingness or language barriers precluding adequate understanding or cooperation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult participants with type 2 diabetes and naive to injectable glucose-lowering treatment.
Sampling Method: Non-Probability Sample
Enrollment: 388 (Actual)
Dates: Start 2023-02-24 (Actual); Primary Completion 2024-06-03 (Actual); Study Completion 2024-06-03 (Actual)

PRIMARY OUTCOMES:
Change in Glycated haemoglobin A1c (HbA1c) | From baseline (week 0) to End of Study visit (V3) (week 34-44)
  Measured as percentage (%)-points.

SECONDARY OUTCOMES:
Relative change in body weight | From baseline (week 0) to End of Study visit (V3) (week 34-44)
  Measured in percentage (%).
Absolute change in body weight | From baseline (week 0) to End of Study visit (V3) (week 34-44)
  Measured in kilogram (kg).
Glycated haemoglobin A1c (HbA1c) less than (<) 7% | At End of Study visit (V3) (week 34-44)
  Measured as Yes or No.
HbA1c reduction greater than or equal to (>=) 1%-points and body weight reduction of greater than or equal to (>=) 5% | From baseline (week 0) to End of Study visit (V3) (week 34-44)
  Measured as Yes or No.
HbA1c reduction greater than or equal to (>=) 1%-points and body weight reduction of greater than or equal to (>=) 3% | From baseline (week 0) to End of Study visit (V3) (week 34-44)
  Measured as Yes or No.

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Transparency dept. 2834, Study Director — Novo Nordisk A/S

IPD SHARING:
Plan to Share IPD: Yes
According to the Novo Nordisk disclosure commitment on novonordisk-trials.com.
URL: http://novonordisk-trials.com

REFERENCES:
- [Derived] Sanyal D, Saboo B, Phatak SR, Kumar PKM, Basu D, Verma N, Nair A, Bhattacharjee K, Aneja P, Makkar BMM, Negalur V, Mithal A, Unnikrishnan AG. Real-World Usage of Once-Daily Oral Semaglutide in Adults with Type 2 Diabetes: Findings from PIONEER REAL India. Indian J Endocrinol Metab. 2025 Sep-Oct;29(5):523-530. doi: 10.4103/ijem.ijem_179_25. Epub 2025 Oct 25. PMID 41229720